CLINICAL TRIAL: NCT06256770
Title: A Trial Study on Evaluation the Safety and Efficacy of Rigid Breathable Scleral Contact Lenses (Model: KTSL ) of Astigmatism,Myopia or Hyperopia
Brief Title: Evaluation of the Safety and Efficacy of Rigid Breathable Scleral Contact Lenses for the Correction of Ametropia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: zhangyi2023
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-02

CONDITIONS: Ocular Surface Disease; Irregular Astigmatism; Contact Lens Complication; Corneal Astigmatism
Keywords: Ocular Surface Disease; Irregular Astigmatism; Contact Lens Complication; Corneal Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- scleral contact lenses group: The selected patients were equipped with scleral contact lenses to evaluate their best corrected visual acuity, refraction, ocular surface condition, and fitting status of contact lenses.
- RGP group: The selected patients were equipped with RGP to evaluate their best corrected visual acuity, refraction, ocular surface condition, and fitting status of contact lenses.

SUMMARY:
To evaluate the short-term efficacy and safety of scleral contact lens in the clinical treatment of patients with irregular astigmatism after corneal transplantation by analyzing ocular parameters and ocular surface conditions of patients after corneal transplantation.

ELIGIBILITY:
Inclusion Criteria:

1.8 ≤ age ≤ 55 years old;2.The diopter of one or both eyes is -25.00~+25.00 D (including -25.00D and +25.00D), and corneal astigmatism caused by any reason (including keratoconus, irregular cornea) ≥0.75D.

Exclusion Criteria:

1.Patients who are judged by the investigator to be unsuitable for corneal endothelial cells;2.Dry eye ;3.Abnormal IOP ;4.Overt strabismus;5.Bacterial, fungal, viral and other active corneal infections;6. Being used may cause dry eyes or affect the eyeball or affect vision or affect the angle drugs such as membrane curvature;7.Corneal sensory, active corneal lesions;8.Conventional slit lamp microscopy and ophthalmoscopy, corneal diseases, iris cyclitis, chronic uveitis, cataract and vitreoretina related eye diseases disease or active and progressive disease;9.Other eye diseases: such as dacryocystitis, eyelid diseases and eyelid abnormalities or infections, eye muscle-related diseases, optic pathway diseases, glaucoma;10.Patients with systemic diseases that cause immunocompromise;History of allergy to contact lenses or contact lens care solution;11.History of allergy to contact lenses or contact lens care solution;12.Pregnant, lactating or planning to become pregnant in the near future;13.Subjects who are considered by the investigator to be unable to wear rigid contact lenses after comprehensively considering the corneal parameters, morphological characteristics and refractive examination results of the examination results;14.Those who have worn hard contact lenses within 30 days or soft hydrophilic contact lenses within 10 days;15.Those who participated in other drug clinical trials 3 months before screening and participated in other medical device clinical trials within 30 days;16.one-eyed patients;17.Those who have a strong sense of foreign body and cannot tolerate it and have poor compliance, and cannot be timely and regular to the medical institution for medical treatment as required;18.Other conditions judged by the investigator that the patient is not suitable for enrollment.

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with corneal astigmatism
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of Best Corrected Vision Acuity | One year
  The percentage of eyes with best corrected visual acuity improved by two lines or more (compared to best corrected visual acuity with glasses) or 5.0 or greater (standard logarithmic visual acuity chart) after 1 month ± 7 days of contact lens wear.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity and Refraction with Contact Lenses | One year
  1. Contact lenses for best corrected visual acuity. List the visual acuity of wearing glasses 7 days±3 days,1 month±7 days, and 3 months±14 days after wearing glasses. To provide the statistical analysis results of spectacle visual acuity in the experimental group and the control group;
  2. Diopter. The diopters of 7 days±3 days,1 month±7 days, and 3 months±14 days after wearing glasses were listed, and the results of diopter analysis in the experimental group and the control group were provided.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Prof, Study Chair — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided